CLINICAL TRIAL: NCT05897086
Title: Nerve Repair Using Hydrophilic Polymers to Improve Tactile and Erogenous Neophallus Sensation
Brief Title: Polyethylene-glycol Assisted Nerve Repair in Phalloplasty
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Wesley Thayer, Professor of Plastic and Reconstructive Surgery, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 221616
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Gender Dysphoria
Keywords: Phalloplasty
MeSH Terms: conditions — Gender Dysphoria | interventions — polyethylene glycol 3350

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention) (No Intervention): For the control groups, epineural repair will be undertaken in the standard end-to-end fashion using interrupted nylon suture after irrigation of the wound with normal saline as deemed necessary by the operating surgeon.
- Experimental (Experimental): For the experimental group, after obtaining hemostasis, prior to neurorrhaphy, the operative field will be irrigated with calcium-free Plasmalyte A® (Baxter: Deerfield, IL) throughout the neurorrhaphy. At this point, the nerves will be repaired using standard suture neurorrhaphy techniques. Subsequently, approximately 1 or 2 drops of 5mg/ml (0.5%) methylene blue in sterile water solution are applied to the trimmed nerve endings. Then, approximately 2 ccs of a 190 mM solution of 50% PEG 3.35 kD in sterile water will be irrigated onto the neurorrhaphy site and the surgeon will wait one minute prior to continuing. Following this, the repaired nerve will be irrigated with calcium-containing Lactated Ringers (Hospira; Lake Forest, IL).
  Interventions: Drug: Polyethylene Glycol 3350

INTERVENTIONS:
Drug: Polyethylene Glycol 3350 — Topical irrigation with approximately 2 ccs of a 190 mM solution of 50% PEG 3.35 kD in sterile water
  Arms: Experimental

SUMMARY:
Phalloplasty, a genitourinary surgery for transmasculine patients, reconstructs a neophallus using tissue transferred from other parts of the body to the groin. However, this technique fails to provide adequate sensation, causing regret and persistent dysphoria. Peripheral nerve regeneration is the greatest barrier to sensory recovery, given the slow rate of regrowth coupled with the negative effects of axonal degeneration. Topical application of polyethylene glycol (PEG) fuses severed axonal membranes, restoring the nerve's immediate ability to conduct electrical signals across the repair site. The investigators hypothesize that utilizing PEG in phalloplasties will significantly improve neophallus sensation and postoperative quality of life.

DETAILED DESCRIPTION:
With more than 1.6 million transgender and nonbinary (TGNB) individuals in the United States, the investigators have witnessed an exponential increase in the number of gender-affirming surgeries performed in the last 2 decades. Of the affirming surgical spectrum, "bottom" genitourinary surgeries remain the most challenging. Specifically, phalloplasty is a masculinizing surgery for neophallus creation using free tissue transfer from other parts of the body and microvascular techniques for nerve and vessel reattachment. In radial forearm free flap (RFFF) phalloplasty, nerves from the forearm are harvested with the flap and sutured to nerves in the groin to provide postoperative sensation in the neophallus. Despite transmasculine patients ranking sensation as one of their top priorities, standard nerve coaptations performed in phalloplasty fail to provide consistent sensation with scarce dedicated research aimed at enhancing neophallus sensory outcomes. Without scientific advances, phalloplasty will remain far from perfect, negatively affecting patients' sexual health, causing dissatisfaction, and increasing the risk of surgical regret and persistent dysphoria.

Peripheral nerve regeneration remains the limiting factor for ideal sensory recovery due to the slow and inconsistent rates of regeneration, and the negative effects of axonal degeneration that occurs post-injury. The investigators advocate for using polyethylene glycol as a "fusogen" to achieve nerve fusion in peripheral nerve coaptations. Polyethylene glycol (PEG) is a hydrophilic compound that enhances the fusion of the lipid bilayer membrane of severed axons, restoring the nerve's immediate ability to conduct electrical signals across the repair site. The investigators have conducted extensive mammalian and preliminary human studies using our novel PEG-fusion protocol for nerve coaptations. In both ex-vivo and in-vivo studies in rats with severed sciatic nerves, PEG-assisted nerve coaptation restored morphological continuity and led to a remarkable early improvement in functional outcomes. In the first human PEG fusion of injured digital nerves performed by our team, the investigators saw rapid nerve recovery and early functional outcomes as early as one week. Based on the investigator's experience with PEG fusion, the investigators will be conducting a randomized clinical trial to test the efficacy of PEG-assisted nerve coaptation in achieving superior neophallus sensory function following phalloplasty.

ELIGIBILITY:
Inclusion Criteria:

* over the age of 18
* preoperative diagnosis of gender dysphoria and present for planned radial forearm free flap phalloplasty
* willing to comply with all aspects of treatment as well as the study evaluation schedule

Exclusion Criteria:

* a known allergy to the study drug
* a hematocrit of 54% or higher
* a history of venous thromboembolism (VTE), peripheral phlebitis, stroke, or myocardial infarction within the last 6 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Transmasculine
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2028-12-30 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Medical Research Council Classification (MRCC) | 15 months
  measures sensory recovery

SECONDARY OUTCOMES:
Vanderbilt Mini-PROM for Gender-Affirming Surgery(VMP-G) | 15 months
  This questionnaire measures psychosocial well-being and resolution of gender-dysphoria
Sexual Functioning and Sensation Questionnaire | 15 months
  measures sexual function and subjective/erogenous sensation

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Thayer, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States